Study Title: Partnering with WIC to Prevent Excessive Weight Gain in Pregnancy

NCT Number: NCT03707834

**Documents Included:** English & Spanish IRB Approved Consents

Date of IRB Approval: 06/18/2023

Temple IRB Approved 06/18/2023

# Consent to Participate in Study – Remote Version

**Title of research:** Partnering with WIC to prevent excessive weight gain in pregnancy (#BabyBeHealthy)

#### Investigator and Department:

Sharon J. Herring, MD, MPH

Associate Professor of Medicine, Clinical Sciences, and Ob/Gyn Lewis Katz School of Medicine at Temple University

Center for Obesity Research and Education

## Why am I being invited to take part in this research?

You are being asked to participate in a research study to find out whether a healthy lifestyle program is an acceptable and effective way for pregnant women to improve their eating and activity, and control their weight gain, compared to usual WIC care. The goal of the program is to enhance the health of African American and Latina women during pregnancy.

We invite you to take part in this research study because you are a WIC participant, self- identify as African American or Latina, are less than 16 weeks' pregnant, and are at least 18 years of age.

#### What should I know about this research?

- Someone will explain this research to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

#### Who can I talk to about this research?

If you have questions, concerns, or complaints, or think the research has hurt you, contact the research team and/or Principal Investigator (Sharon J. Herring, MD, MPH) by phone at (215) 707-2234 or by mail at 3223 N. Broad Street, Suite 175, Philadelphia, PA, 19140. This research has been reviewed and approved by an Institutional Review Board. You may talk to them at (215) 707-3390 or e-mail them at: irb@temple.edu for any of the following:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# Why is this research being done?

Both eating unhealthy and limited physical activity during pregnancy are linked to higher rates of obesity, diabetes, and heart disease for mothers and their babies. We are doing this research to find out if using text messages and social media paired with counseling in the WIC setting will help improve mothers' eating, activity, and weight control in pregnancy. If the answer is yes, our research may lead to substantial improvements in the health of mothers with young children.

### How long will I be in this research?

We expect that you will be in this research for approximately 18 months after your enrollment.

## What happens if I agree to be in this research?

Once enrolled, you will be randomly assigned (like the flip of a coin) to one of 2 groups (the Healthy Lifestyle Group or Usual WIC Care). This means that you do not have a choice in which group you are put into. The treatment you get will be chosen by chance, like flipping a coin. Neither you nor the study team will choose what treatment you get. You will have a 50/50 chance of being in either group.

#### **PROCEDURES**

If you are in the <u>Healthy Lifestyle Group</u>, you will get information and strategies to help you eat healthier and be more active during pregnancy.

The healthy lifestyle program will last approximately 24 weeks (from early pregnancy through delivery). You will receive daily text messages with tips and video links about staying healthy in pregnancy along with reminder texts to monitor your eating and activity goals. You will additionally have monthly to bimonthly study-related phone calls from a WIC nutritionist to set goals, overcome challenges, and give you new information about diet and activity while you're in the program. These calls will last 15- 30 minutes and will be audiotaped. An optional private Facebook group and an optional private Instagram profile will be available as well, where you can interact with other mothers in the study and learn new tips about staying healthy.

Once you deliver your baby, you will no longer receive text messages, telephone calls, or study-related social media posts about eating and activity. However, you will remain in the study until your baby is 1 year of age.

If you are in the <u>Usual WIC Care Group</u>, you will receive usual advice about nutrition and activity during pregnancy from WIC along with some additional handouts from The American College of Obstetricians and Gynecologists.

#### MEDICAL SCREENING

In order to participate in this study, your medical chart will be reviewed by our study physician (Sharon J. Herring, MD, MPH) for any medical exclusions, including medical conditions and/or medications that could potentially influence nutrition and weight gain in pregnancy (such as bariatric surgery, stroke, frequent seizures, HIV, thyroid disease, pre-existing diabetes, gallbladder disease, cardiovascular disease, substance abuse, current use of risperidone, quetiapine, olanzapine, phentermine, etc.).

#### **ASSESSMENTS**

We will ask you some questions about your past medical history by phone to make sure you are

eligible to participate in the study. If you are eligible, you will schedule a combined CORE Screening and Enrollment call where you will consent to participate. We will ask you to selfreport your weight and height, ask you to complete a number of questionnaires to learn information about your lifestyle, including your previous 24-hour food intake, and verify that you meet all inclusion criteria. After completion of all questionnaires, you will be officially enrolled and randomly assigned to either the Healthy Lifestyle Group or Usual WIC Care Group. We will then send you a BodyTrace scale to use for your weight at each time point. We will conduct follow-up phone calls at 36-38 weeks' of pregnancy (end of pregnancy), 6 months postpartum, and 12 months postpartum and complete questionnaires similar to your CORE Screening/Enrollment call. If you agree, at your 6 month and 12 month postpartum calls, we will additionally have you sign medical record release forms to get your baby's weight and length. Each of these calls will last approximately 45 to 60 minutes and will be scheduled ahead of time. If public health guidelines allow and you consent, these calls may be conducted as in-person visits at Temple's CORE office (3223 N. Broad Street, Suite 175) or if transportation is an issue, we will conduct these visits at your home. A detailed study timetable and list of all procedures at each visit are shown below:

| | | Time point | | | |
|---|---|---|---|---|---|
| Measure | Phone<br>Screening | CORE<br>Screening/<br>Enrollment | 36-week<br>GA | 6-Mo<br>Postpartum | 12-Mo<br>Postpartum |
| | | Baseline | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| Screening Eligibility Form | X | | | | |
| Informed Consent | | Х | | | |
| Questionnaires | | Х | Х | Х | X |
| Maternal Weight | | X | Х | Χ | X |
| Maternal Height | | Х | X | Χ | X |
| Infant Weight | | | | Χ | X |
| Infant Length | | | | Χ | X |
| 24-Hour Recall of Food Intake | | Х | X | | |
| Maternal Medical Record Review | | Х | X | Χ | X |
| WIC Medical Record Review | | Х | Х | Χ | X |

# What other choices do I have besides taking part in this research?

There are several methods of improving nutrition and activity during pregnancy that do not require the methods described in this program. Sharon Herring, MD, MPH, or one of her associates, will provide suggestions for alternative methods if you do not wish to participate in this study.

## Is there any way being in this research could be bad for me?

There is minimal risk to both you and your baby during pregnancy - you will be encouraged to participate in moderate physical activity (walking) and eating behaviors that are associated with the best outcomes for mother and baby. Recommendations for physical activity and nutrition will not differ from established public health recommendations. There is a small risk of muscle sprains, other soft tissue injuries, or bone injuries from exercise; however, you will be given information about proper stretching and the importance of a warm-up and cool-down period to minimize injury. You should contact your obstetrician for any health concerns.

You may become uncomfortable when talking about your height or weight. To minimize discomfort, all staff will conduct phone calls from a private space to ensure all of your information

is kept confidential. Additionally, you may become uncomfortable answering questions (e.g., about demographics, dietary intake, or health-related quality of life). To minimize discomfort by participants, all staff members have experience interacting with pregnant women. Data will only be labeled with an identification number (no names) and only appropriate research staff will have access to this number

In addition, there is a small risk of loss of privacy due to the Facebook group and/or Instagram profile. All healthy lifestyle participants have three different options for the manner in which they join the Facebook group, each corresponding to the level of privacy they wish to have: Option 1) Participants can choose to link their own existing private Facebook account with the private Facebook group, allowing other participants to see all of the content on their individual Facebook page; Option 2) Participants can choose to link their own existing private Facebook account with restrictions to the private Facebook group, allowing other participants to see only the content on their individual Facebook pages that they permit them to view; Option 3) Participants can choose to create an alias Facebook account exclusively for joining the Healthy Lifestyle Group, prohibiting the other participants from accessing any of the content on the individual Facebook pages that they maintain for personal, private use. For Instagram, there are two options: Option 1) Participants can use their own existing Instagram profile to follow the private study Instagram profile: Option 2) Participants can choose to create an alias Instagram account exclusively for following the study Instagram profile, prohibiting other participants from accessing any of the content on their individual Instagram profile that they maintain for personal, private use. Study staff will review and respond to any comments made or messages sent on both social media platforms to dispel misinformation, provide support, and monitor progress, distress and/or side effects from the program.

### Will being in this research help me in any way?

Participation in the program may benefit you in several ways. First, the program may result in improvements in your eating and activity, which may be associated with resolution/improvements in medical conditions made worse by poor diet or excess weight (e.g., diabetes, high blood pressure). In addition, your progress and health will be monitored throughout the program and results of the assessments will be made available to you to share with your doctor.

However, you cannot be guaranteed any medical benefit from participating in this study. No one can predict beforehand whether you will respond favorably to the treatment provided and, thus, experience improvements in your health.

The anticipated benefits to society are great, as the information developed for this study may help other mothers in the future.

# What happens to the information collected for this research?

To the extent allowed by law, we limit the viewing of your personal information to people who have to review it. We cannot promise complete secrecy. The IRB, Temple University, Temple University Health System, Inc. and its affiliates, and other representatives of these organizations may inspect and copy your information.

We will communicate with you by text message. In the Healthy Lifestyle Group, we will also communicate with you by phone and we will ask you to weigh yourself on a cellular- connected scale. To send and receive phone calls and text messages, and to store your study information and weights, we use companies such as Twilio, Google Cloud Platform, and BodyTrace. These companies will take measures to keep information safe on their servers (such as keeping the data

When we talk to you on the phone, we will speak with you from a private space.

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

If you choose to participate, we will ask you to sign an Authorization to Release/Obtain Information for the purpose of collecting your prenatal and delivery records. Medical records will be requested and collected by study staff via HelloFax, a secured and encrypted online fax service and stored at CORE on a HIPAA-compliant file server.

Federal law provides additional protections of your personal information. These are described in an attached document titled "Authorization to use and disclose your protected health information".

#### What will I be paid for taking part in this research?

If you agree to take part in this research, you will receive \$100 after completing all CORE Screening/Enrollment questionnaires and being officially enrolled (to reimburse participants for time). All enrolled participants will also receive a diaper bag and a scale to weigh themselves at each study time point after their CORE Screening/Enrollment call; mothers in the intervention group will additionally have a scale, water bottle, measuring bowls, cookbook and healthy snacks included in their bag. Enrolled participants will additionally receive \$75 after completion of their 36- week gestation call, and \$50 after completion of their 6-month postpartum and 12-month follow-up calls.

Total compensation for completing all assessments will be \$275.00 (for both groups). You will either be texted or emailed VISA e-gift cards (preferred method) or mailed plastic VISA gift cards at the end of each visit. If you are randomized to the Healthy Lifestyle Group, you will be eligible to win a monthly raffle prize. The prizes will vary each month and are valued between \$75 and \$100. You will receive 1 raffle entry for each monitoring text you send. Monthly raffles will be held (run by study staff) on the last day of every month and winners will be contacted via text message.

Federal tax law requires to you to report this payment as income to the Internal Revenue Service.

You may be asked to tell us your social security number. If payments are more than \$599.00, we will report them to the Internal Revenue Service and send you a Form 1099-MISC. If you do not give us your social security number, you may take part in this research if you agree to not be paid.

this study.

## **Optional Permissions Requested**

#### 1. Permission to audiotape

2.

If you are in the Healthy Lifestyle Group, we request permission to audiotape your study-related WIC nutritionist phone calls. These audiotape recordings will be used as part of your treatment and for training. Please know that you can withdraw your permission at any time without prejudice to you or your relationship with the study, Temple University, WIC, or the Study doctor and team.

| or the St | udy doctor and team. |
|---|---|
| | Yes, I give permission for my study-related WIC phone calls to be audiotaped. |
| | No, I do not give permission for my study-related WIC phone calls to be audiotaped. |
| We are a<br>at 6-mor<br>signature | sion for infant measures asking permission to request the weights and lengths from your infant's pediatrician of this and 1-year of age. An additional Medical Record Release form will be sent for e. We are interested in this information so we can learn if the program also has an n your infant. |
| | Yes, I give permission to have my infant's weight and length measured for this study. |
| | No, I do not give permission to have my infant's weight and length measured for |

#### 3. Permission for in-person assessments contingent upon access to an effective Covid-19 vaccine

We are asking permission to conduct the below assessments once there is access to an effective vaccine for Covid-19 and the risk of transmission to participants significantly drops, therefore, allowing in-person visits to resume.

| Assessment | Yes | No | Participant<br>Initials |
|---|---|---|---|
| Maternal Height and Weight: Measure height and weight at all inperson visits. | | | |
| <u>Maternal Blood Pressure</u> : Perform blood pressure at all in-person visits. | | | |
| GT3X device: You will be given a GT3X+ wrist actigraph for measuring physical activity for approximately 7 days. Activity will be monitored at enrollment and end-of-pregnancy. | | | |
| Infant Length and Weight: Measure your infants' length and weight at your 6-month and 12-month postpartum visits. | | | |
| Study related progress reports: If you are in the Healthy Lifestyle Group, we request permission to put a printed copy of your #BabyBeHealthy progress report in your WIC chart once in-person WIC visits resume. | | | |

| Your signature documents your permission to take part in this research. | |
|---|---|
| Signature of subject | Date |
| Printed name of subject | - |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | - |

**Temple IRB Approved** 

06/18/2023

## Consentimiento para Participar en el Estudio - Versión Remota

**Titulo de la investigación:** Asociándose con WIC para prevenir el aumento de peso excesivo en el embarazo (#BebéSeaSaludable)

## Investigadora y Departmento:

Sharon J. Herring, MD, MPH

Profesora Asociada de Medicina, Ciencias Clínicas y Ginecólogo Obstetra (Ob / Gyn) Escuela de Medicina de Lewis Katz en la Universidad de Temple

Centro de Investigación y Educación de Obesidad (CORE)

## ¿Por qué se me invita a participar en esta investigación?

Se le pide que participe en un estudio de investigación para averiguar si un programa de estilo de vida saludable es una forma aceptable y efectiva para que las mujeres embarazadas mejoren su alimentación y actividad, y controlen su aumento de peso, en comparación con el cuidado usual de WIC. El objetivo del programa es mejorar la salud de las mujeres Latinas y Afro-Americanas durante el embarazo.

Le invitamos a participar en este estudio de investigación por que eres una participante de WIC, se auto-identifica como Latina o Afro-Americana, tiene menos de 16 semanas de embarazo, y tiene por lo menos 18 años de edad.

## ¿ Qué debo saber acerca de esta investigación?

- Alguien le explicará esta investiagción.
- La decisión de participar o no participar es suya.
- Puede optar por no participar en el estudio.
- Puede aceptar participar y cambiar su decisión en el futuro.
- Su decisión al respecto no se considerará en su contra.
- Puede hacer todas las preguntas que desee antes de tomar una decisión.

# ¿Con quien puedo hablar acerca de esta investigación?

Si tiene preguntas, inquietudes o quejas, o cree que la investigación le ha provocado algún daño, póngase en contacto con el equipo de investigación o la investigadora principal (Sharon J. Herring, MD, MPH) por teléfono al (215) 707-2234 o por correo a 3223 N. Broad Street, Suite 175, Filadelfia, PA, 19140. Esta investigación ha sido revisada y aprobada por un Comité de Revisión Institucional. Puede comunicarse con dicho comité llamando al (215) 707-3390 o por correo electronico: irb@temple.edu por cualquiera de los siguientes motivos:

- Sus preguntas, inquietudes o quejas no estan siendo contestadas por el equipo de investigación.
- Usted no puede comunicarse con el equipo de investigación.

- Usted quieres hablar con alguien que no sea el equipo de investigación.
- Usted tiene preguntas sobre sus derechos como un sujeto de investigación.
- Usted desea obtener información o proporcionar informacion sobre esta investigación.

## ¿Por qué se realiza esta investiagción?

Comer poco saludable y hacer actividad fisica limitada durante el embarazo están relacionados con riesgos de salud más altas de obesidad, diabetes y enfermedades del corazón para las madres y sus bebés. Estamos haciendo esta investigación para averiguar si usando mensajes de texto y las redes sociales combinado con consejería de nutricion en el centro de WIC ayudará a mejorar la alimentación, la actividad y el control de peso de las madres durante el embarazo. Si la respuesta es Si, nuestra investigación puede llevar a mejores resultados en la salud de las madres con niños pequeños.

## ¿Cuánto tiempo participaré en esta investigacion?

Esperamos que usted participe en esta investigación por aproximadamente 18 meses después de su inscripción.

# ¿ Qué sucede si acepto participar en esta investigación?

Cuando este inscrita en el estudio, se le asignará al azar a participar (como si fuera al seleccionar cara o cruz en una moneda) en uno de los 2 grupos (el Grupo de Estilo de Vida Saludable o cuidado usual de WIC). Esto significa que no tienes una opción en qué grupo se le asigna. El tratamiento que recibas será elegido al azar, como tirar una moneda. Ni usted ni el equipo del estudio elegirán el tratamiento que recibirá. Tendrá una probabilidad de 50/50 de estar en cualquiera de los grupos.

#### **PROCEDIMIENTOS**

Si está en el <u>Grupo de Estilo de Vida Saludable</u>, conseguirás información y estrategias para ayudarla a comer más saludable y ser más activa durante el embarazo.

El programa de estilo de vida durará aproximadamente 24 semanas (desde el embarazo temprano hasta el parto de su bebé). Recibirás mensajes de texto diarios con consejos y videos sobre cómo mantenerse saludable durante el embarazo. Junto con textos recordatorios para monitorear sus metas de alimentación y actividad. Además, recibirá llamadas telefónicas mensuales a llamadas bimensuales relacionadas con el estudio con una nutricionista de WIC para establecer metas, superar los desafíos, y le dará nueva información sobre la dieta y la actividad mientras está en el programa. Estas llamadas durarán entre 15 y 30 minutos y serán grabadas en audio. También estará disponible un grupo privado de Facebook opcional y un perfil privado de Instagram opcional, donde podrá interactuar con otras madres en el estudio y aprender nuevos consejos sobre cómo mantenerse saludable.

Una vez despues del parto de su bebé, ya no recibirá mensajes de texto, llamadas telefónicas, ni publicaciones en redes sociales relacionadas con el estudio sobre alimentación y actividad. Sin embargo, permanecerá en el estudio hasta que su bebé tenga 1 año de edad. Si está en el Grupo de Cuidado Usual de WIC, recibirá consejos sobre nutrición y actividad durante el embarazo de parte de WIC junto con algunos folletos adicionales del Colegio Americano de Obstetras y Ginecólogos.

#### REVISIÓN DE INFORMACIÓN MÉDICA

Para poder participar en este estudio, su record/registro medico (información médica) sera revisado por nuestro médico del estudio (Sharon J. Herring, MD, MPH), el medico revisará su historial medico para cualquier exclusión médica, incluso condiciones médicas y / o medicamentos que podrían influir la nutrición y el aumento de peso durante el embarazo (como cirugía bariátrica, derrame cerebral, convulsiones frecuentes, VIH, enfermedad de la tiroides, diabetes pre-existente, enfermedad de la vesícula biliar, enfermedad cardiovascular, abuso de sustancias, uso actual de risperidone, quetiapine, olanzapine, phentermine, etc.).

#### **EVALUACIÓNES**

Le haremos algunas preguntas sobre su historial médico anterior por teléfono para asegurarnos que usted eres elegible para participar en el estudio. Si eres elegible, usted programará una llamada para realizar su evaluación combinada de la Evaluación de Elegibilidad e Inscripción de CORE donde consentirás participar en el estudio. Le pediremos que autoinforme su peso y estatura, le pediremos que complete una serie de cuestionarios para obtener información sobre su estilo de vida, incluyendo su registro de la ingesta de alimentos de las 24 horas anteriores y verificaremos que usted cumple con todos los requisitos de inclusion. Después de completar todas los cuestionarios, se inscribirá oficialmente en el estudio y se le asignará al azar al Grupo de Estilo de Vida Saludable o el grupo de Cuidado Usual de WIC. Luego le enviaremos una báscula de BodyTrace para que usted mida su peso en cada punto de tiempo. Realizaremos llamada telefonicas de seguimiento a las 36-38 semanas de embarazo (final del embarazo), 6 meses después del parto y 12 meses después del parto y completará cuestionarios similares a su llamada de Evaluación de Elegibilidad/Inscripción. Si está de acuerdo, en sus llamadas de 6 meses y 12 meses posparto, también mediremos el peso y la longitud de su bebé. Cada una de estas llamadas durará aproximadamente 45 a 60 minutos y se programará con anticipación. Si las pautas de salud pública lo permiten y usted da su consentimiento, estas llamadas pueden realizarse como visitas en persona en la oficina de CORE en Temple (3223 N. Broad Street, Suite 175) o si el transporte es un problema, haremos estas visitas en su hogar. A continuación se muestra un calendario detallado del estudio y una lista de todos los procedimientos en cada visita:

| | | Punto de Tiempo | | | |
|---|---|---|---|---|---|
| Medida | Evaluación<br>de<br>Elegibilidad<br>por<br>Telefono | Evaluación<br>de<br>Elegibilidad/<br>Inscripción<br>de CORE | 36 Semanas<br>EG | 6 Meses<br>Posparto | 12 Meses<br>Posparto |
| | | Inicial | Seguimiento 1 | Seguimiento 2 | Seguimiento 3 |
| Formulario de Evaluación de Elegibilidad | Х | | | | |
| Consentimiento<br>Informado | | Х | | | |
| Cuestionarios | | X | X | X | X |
| Peso Materno | | X | X | X | X |
| Estatura Materna | | X | X | X | X |
| Peso Infantil | | | | X | X |

| Longitud Infantil | | | Х | Х |
|-------------------------|---|---|---|---|
| Registros de Ingesta de | | | | |
| Alimentos de las | | | | |
| Ultimas 24 Horas | X | X | | |
| (ASA-24) | | | | |
| Revisión de | | | | |
| Registros Médicos | | | | |
| (información médica) | X | Χ | X | X |
| Maternos | | | | |
| Revisión de Registros | | | | |
| Médicos de WIC | X | X | X | X |

# ¿Qué otras opciones tengo, además de tomar parte en esta investigación?

Hay varios métodos para mejorar la nutrición y la actividad durante el embarazo que no requieren los métodos descritos en este programa. Sharon Herring, MD, MPH, o uno de sus asociados, proporcionará sugerencias sobre métodos alternativos si no desea participar en este estudio.

# ¿Hay alguna forma de estar en esta investigación que podría ser malo para mí?

Existe un riesgo mínimo tanto para usted como para su bebé durante el embarazo: sera animada a participar en actividades físicas moderadas (caminar) y implementar hábitos alimenticios asociadas con los mejores resultados para la madre y el bebé. Las recomendaciones para la actividad física y la nutrición no serán diferentes de las recomendaciones establecidas por la salud pública. Existe un pequeño riesgo de esguinces musculares, otras heridas de tejidos blandos o heridas de hueso por el ejercicio; sin embargo, se le dará información sobre el estiramiento adecuado y la importancia de un período de calentamiento y enfriamiento para minimizar las heridas. Debe ponerse en contacto con su obstetra para cualquier problema o preocupación de salud.

Puede sentirse incómoda al hablar de su estatura o peso. Para minimizar la incómodidad, todo el personal del estudio realizará llamadas telefónicas desde un espacio privado para garantizar que toda su información se mantenga confidencial. Además, puede sentirse incómoda al responder preguntas (por ejemplo, sobre datos demográficos, ingesta dietética o calidad de vida relacionada con la salud). Para minimizar la incómodidad de los participantes, todos los miembros del personal tienen experiencia interactuando con mujeres embarazadas. Los datos solo se identificaran con un número de identificación (sin nombres) y solo el personal de investigación apropiado tendrá acceso a este número.

Además, existe un pequeño riesgo de pérdida de privacidad debido al grupo de Facebook y / o perfil de Instagram. Todas las participantes del estudio tienen dos opciones diferentes para la forma en que se unen a la página, cada uno correspondiente al nivel de privacidad que desean tener: Opción 1) Las participantes pueden elegir enlazar su propia cuenta privada existente de Facebook con el grupo privado de Facebook del estudio,permitiendo a las otras participantes ver todo el contenido en su página de Facebook individual; Opción 2) Las participantes pueden optar por enlazar sus propias cuentas privadas de Facebook con restricciones al grupo privado de Facebook, permitiendo a otras participantes ver solo el contenido de sus páginas individuales de Facebook que les permiten ver; Opción 3) Las participantes pueden optar por crear una cuenta de alias en Facebook exclusivamente para unirse al Grupo de Estilo de Vida Saludable,

prohibiendo a las otras participantes el acceso a cualquiera de los contenidos en las páginas individuales de Facebook que mantienen para uso personal o privado. Para Instagram, hay dos opciones: Opción 1) Las participantes pueden usar su propio perfil de Instagram existente para seguir el perfil de Instagram del estudio privado; Opción 2) Las participantes pueden optar por crear una cuenta de alias en Instagram exclusivamente para seguir el perfil de Instagram del estudio, prohibiendo que otras participantes accedan el contenido de su perfil de Instagram individual que mantienen para uso personal y privado. El personal del estudio revisará y responderá a cualquier commentario o mensaje enviado en ambas plataformas de redes sociales para disipar información errónea, dar apoyo y monitorear el progreso, la angustia y / o los efectos secundarios del programa.

### ¿Me ayudará de alguna manera participar en esta investigación?

La participación en el programa puede beneficiarla de varias maneras. Primero, el programa puede dar mejor resultados en su alimentación y actividad, que pueden estar asociadas con la resolución / mejoramiento en condiciones médicas empeoradas por una dieta poco saludable o un exceso de peso (por ejemplo, diabetes, presión arterial alta).

Además, su progreso y su salud se controlarán durante todo el programa y los resultados de las evaluaciones se pondrán a su disposición para compartir con su médico. Sin embargo, no se le puede garantizar ningún beneficio médico por participar en este estudio. Nadie puede predecir de antemano si usted responderá favorablemente al tratamiento proporcionado y asi, si resultara en mejore resultados de su salud.

Los beneficios anticipados para la sociedad son excelentes, ya que la información desarrollada para este estudio puede ayudar a otras madres en el futuro.

# ¿Que occure con la información recolectada para esta investigación?

En la medida permitida por la ley, limitamos la visualizacion de su información personal a las personas que tienen que revisarlas. No podemos prometer una confidencialidad completa. El Comité de Revisión Institucional (IRB), Universidad de Temple, El Systema de Salud de la Universidad de Temple, Inc. y sus filiales, y otros representantes de estas organizaciones, pueden inspeccionar y copiar su información.

Nos comunicaremos con usted por mensaje de texto. En el Grupo de Estilo de Vida Saludable, también nos comunicaremos con usted por teléfono y le pediremos que se pese en una bascula de peso conectada por un servicio celular. Para enviar y recibir llamadas telefónicas y mensajes de texto, y para guardar su información del estudio y su peso, utilizamos compañías como Twilio, Heroku, Plataforma de Google Cloud, y BodyTrace. Estas compañías tomarán medidas para mantener la información segura en sus servidores (como mantener los datos encriptados), pero ningún sistema es completamente seguro.

Cuando hablemos con usted por teléfono, lo haremos en un espacio privado. Podemos publicar los resultados de esta investigación. Sin embargo, mantendremos su nombre y otra información de identificación confidencial.

La descripción de este ensayo clínico estará disponible en http://www.ClinicalTrials.gov, según lo exige la ley de EE. UU. Este sitio web no incluirá información quregiste pueda identificarla. A lo sumo, el sitio web incluirá un resumen de los resultados. Puede buscar en este sitio web en

cualquier momento.

Si elige participar, le pediremos que firme una autorización para divulgar / obtener información con el fin de recolectar sus records/registros prenatales y del parto. Los records/registros médicos serán solicitados y recolectados por el personal del estudio a través de HelloFax, un servicio de fax en línea seguro y cifrado, y almacenados en el departamento de CORE en un servidor de archivos compatible con HIPAA.

La ley federal proporciona protecciones adicionales de su información personal. Estos se describen en un documento adjunto titulado "Autorización para usar y divulgar su información médica protegida".

### ¿ Qué me pagarán por participar en esta investigación?

Si acepta participar en esta investigación, recibirá \$100 despues de completar todo los cuestionarios de la Evaluación de Elegibilidad e Inscripción de CORE y estar inscrita oficialmente (para reembolsar a las participantes por tiempo). Las participantes inscritas en el estudio también recibirán una bolsa de pañales y una báscula para pesarse en cada punto de tiempo del estudio después de su evaluación de elegbilidad e inscripción de CORE; las madres en el grupo de intervención tendrán adicionalmente una báscula de peso, un envase de agua, tazas de medir porciónes,un libro de recetas, y meriendas saludable incluidos en su bolsa. Las participantes inscritas en el estudio recibirán \$75 adicional despues de completar su visita de gestación de 36 semanas y \$50 después de completar sus llamadas de seguimiento de 6 meses y 12 meses posparto.

La compensación total por completar todas las evaluaciones será \$275.00 (para ambos grupos). Las tarjetas de regalo VISA electrónicas se enviarán a usted por mensaje de texto o correo electrónico (metodo preferido) o se enviarán tarjetas plasticas de regalo VISA al final de cada visita por correro. Si eres asignada al Grupo de Estilo de Vida Saludable, también serás elegible para ganar un premio de la rifa mensual. Los premios variarán cada mes y se valoran entre \$75 y \$100. Recibirá 1 entrada de la rifa por cada texto de monitoreo que envíe. Las rifas mensuales se harán (a cargo del personal del estudio) el último día de cada mes y las ganadoras serán contactadas por mensaje de texto.

La ley fiscal federal requiere que usted reporte este pago como ingreso al Servicio de Impuestos Internos. Se le puede pedir que nos diga su número de seguro social. Si los pagos superan mas de \$ 599.00, los informaremos al Servicio de Impuestos Internos y le enviaremos un Formulario 1099-MISC. Si no nos proporciona su número de seguro social, puede participar en esta investigación si acepta no recibir un pago.

## Permisos Opcionales Solicitados

#### 1. Permiso para grabar audio

2.

Si estas asignada al Grupo de Estilo de Vida Saludable, solicitamos permiso para grabar en audio las llamadas telefónicas relacionadas con el estudio con la nutricionista de WIC. Estas grabaciones de audio se utilizarán como parte de su tratamiento y para el etrenamiento de nutricionistas de WIC. Por favor tenga en cuenta que puede retirar su permiso en cualquier momento sin perjuicio de usted o su relación con el estudio, la Universidad de Temple, WIC o el equipo y el médico del estudio.

| | SI, yo doy permiso para que las llamadas telefonicas relacionadas con el estudio con la nutricionista de WIC sean grabadas en audio. |
|---|---|
| | _No, no doy permiso para que las llamadas telefónicas relacionadas con el estudio cor<br>la nutricionista de WIC estudio sean grabadas en audio. |
| Estam<br>los 6 n<br>médico | so para tomar las medidas infatiles os pidiendo permiso parapara solicitar los pesos y longitudes al pediatra de su infante a neses y al año de edad. Se enviará un formulario adicional de divulgación de registros os para su firma. Estamos interesados en esta información para que podamos saber si grama también tiene un impacto en su infante. |
| | _Sí, yo doy permiso para medir el peso y la longitud de mi infante para este estudio. |
| | No, no doy permiso para medir el peso y la longitud de mi infante para este estudio. |

# 3. Permiso para realizar evaluaciones en persona contingente al acceso a una vacuna Covid-19 efectiva

Solicitamos permiso para realizar las siguientes evaluaciones una vez que haya acceso a una vacuna eficaz para el Covid-19 y el riesgo de transmisión a los participantes disminuya significativamente, por lo tanto, se permite la reanudación de las visitas en persona.

| | Si | No | Iniciales de la<br>Participante |
|---|---|---|---|
| Estatura y Peso Materna: Medir la estatura y el peso en | | | |
| todas las visitas en persona. | | | |
| Presión Arterial Materna: Realice la presión arterial en | | | |
| todas las visitas en persona. | | | |
| <b>Dispositivo GT3X</b> : Se le entregará un actígrafo de muñeca | | | |
| de GT3X + para medir la actividad física durante | | | |
| aproximadamente 7 días. La actividad será monitoreada al | | | |
| momento de la inscripción y al final del embarazo. | | | |
| Longitud y Peso del Infante: Mida la longitud y el peso de | | | |
| su infante en sus visitas posparto a los 6 y 12 meses. | | | |
| Reportes de Progreso Relacionados con el Estudio: Si | | | |
| está en el Grupo de Estilo de Vida Saludable, solicitamos | | | |
| permiso para poner una copia impresa de su reporte de | | | |
| progreso #BabyBeHealthy en su registro de WIC una vez | | | |
| que se reanuden las visitas de WIC en persona. | | | |

## Bloque de Firmas para Sujetos Adultos con Capacidad de Consentimiento

| Su firma documenta su permiso para participar en esta investigación. | |
|---|---|
| Firma del Sujeto | Fecha |
| Nombre impreso del Sujeto | |
| Firma de la persona que obtiene el consentimiento | Fecha |
| Nombre en letra de imprenta de la persona que obtiene el consentimiento | |